CLINICAL TRIAL: NCT05953337
Title: Radioembolization Oncology Trial Utilizing Transarterial Eye90 (ROUTE 90) for the Treatment of Hepatocellular Carcinoma (HCC)
Brief Title: Radioembolization Trial Utilizing Eye90 Microspheres™ for the Treatment of Hepatocellular Carcinoma (HCC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ABK Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABK-CA-PROT-85
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Carcinoma Non-resectable; Liver Cancer
Keywords: Hepatocellular Carcinoma; Liver Cancer; Liver Diseases; Internal radiation brachytherapy; Radioembolization; Y90; Yttrium-90; Eye90 microspheres
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- EYE90 Microspheres Treatment (Experimental): Radioembolization with Eye90 Microspheres
  Interventions: Device: EYE90 Microspheres Treatment

INTERVENTIONS:
Device: EYE90 Microspheres Treatment — Y90 glass microspheres

SUMMARY:
This is a prospective, multi-center, open-label study to evaluate the effectiveness and safety of Eye90 microspheres® in the treatment of subjects with unresectable Hepatocellular Carcinoma (HCC). Eye90 microspheres is a medical device containing yttrium-90 (Y-90), a radioactive material, and provides local radiation brachytherapy for the treatment of liver tumors.

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of HCC by imaging confirmation with Liver Imaging Reporting and Data System (LIRADS) category 5 or confirmation of HCC via biopsy.
* No extra hepatic disease.
* Up to 3 lesions with at least one lesion ≥ 2 cm in diameter (long axis) measurable by computed tomography (CT), CBCT, or MRI. At least one lesion must be identified as a target lesion as defined by mRECIST.
* Maximal single lesion size of ≤ 8 cm and sum of the maximal tumor dimensions of ≤ 12 cm with the entire tumor burden expected to be treatable within the perfused volume.
* Intent to treat all lesions within a single session.
* Hypervascular on CBCT, CT, or MRI.
* Evidence that > 33% of the total liver volume is disease-free and will be spared Eye90 treatment.
* Life expectancy of ≥ 6 months.
* ≥ 18 years old at the time of informed consent

Exclusion Criteria:

* Platelet count <50,000/microliter or prothrombin (PT) activity > 50% normal.
* Hemoglobin ≤ 8.5 g/dL (subjects that are non-responders to transfusion or medical management must be excluded).
* INR > 1.7 (if anticoagulated, reversal must be achieved prior to any angiographic procedures).
* ALT > 5x upper limit.
* AST > 5x upper limit.
* Bilirubin ≥ 2.0 mg/dL.
* eGFR ≤ 50 mL/min/BSA.
* Macrovascular invasion.
* Incompetent biliary duct system, prior biliary intervention, or a compromised Ampulla of Vater.
* Estimated lung dose > 30 Gy as calculated using the lung shunt fraction and partition model.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 6 months
  The percentage of subjects with ORR using local mRECIST, as assessed by independent panel review.
Duration of response (DoR) | 6 months
  DoR is defined as response ≥ 6 months for ≥ 60% of responders first occurrence of CR or PR
Incidence of adverse events (AEs) | 12 months
  Incidence of AEs, grouped by System Organ Class (SOC) and Preferred Term (PT), relatedness to study treatment/procedure, and severity.
Incidence of serious adverse events (SAEs) | 12 months
  Incidence of SAEs, grouped by SOC and PT, relatedness to study treatment/procedure, and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kennedy, MD, Principal Investigator — Director, Radiation Oncology Research at Sarah Cannon; Ammar Sarwar, MD, Principal Investigator — Director of Radiation Oncology Research, Beth Israel Deaconess Medical Center; Aravind Arepally, MD, Study Director — ABK Biomedical, Inc
Locations (22):
- United States (21):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - University of California - Irvine, Orange, California
  - AdventHealth Radiation Oncology at Altamonte Springs, Altamonte Springs, Florida
  - Miami Cardiac and Vascular Institute at Baptist Hospital Miami, Miami, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Northwestern University Memorial Hospital, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - University of Iowa Health Care, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Beth Israel Deaconess, Boston, Massachusetts
  - University of Missouri - Ellis Fischel Cancer Center, Columbia, Missouri
  - SSM Health Saint Louis University, St Louis, Missouri
  - Weill Cornell Medicine-New York Presbyterian Hospital, New York, New York
  - Charlotte Radiology, Charlotte, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - HCA Healthcare Research Institute (Sarah Cannon), Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Inland Imaging, Spokane, Washington
  - Froedtert Hospital/Medical College of Wisconsin, Milwaukee, Wisconsin
- Vancouver Coastal Health Research Institution (VCHRI), Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No